CLINICAL TRIAL: NCT01969643
Title: A Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety and Tolerability of SGN-LIV1A in Patients With Metastatic Breast Cancer
Brief Title: A Safety Study of SGN-LIV1A in Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNLVA-001
Record Dates: First submitted 2013-10-21; First posted 2013-10-25 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: HER2 Positive Breast Neoplasms; Hormone Receptor Positive Breast Neoplasms; Triple Negative Breast Neoplasms; HER2 Mutations Breast Neoplasms
Keywords: Monomethyl auristatin E; Antibody-drug conjugate; Drug therapy; Metastatic; LIV-1 protein, human; Trastuzumab; Ladiratuzumab vedotin; hLIV22-vcMMAE; Seattle Genetics
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — SGN-LIV1A; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LV Dose Escalation (Experimental)
  Interventions: Drug: ladiratuzumab vedotin
- LV + Trastuzumab (Experimental)
  Interventions: Drug: ladiratuzumab vedotin; Drug: Trastuzumab
- LV Monotherapy (Experimental): LV will be given at the recommended dose (at or below the monotherapy MTD determined in the LV dose escalation arm).
  Interventions: Drug: ladiratuzumab vedotin

INTERVENTIONS:
Drug: ladiratuzumab vedotin — LV will be given into the vein (IV; intravenously)
  Other Names: LV; SGN-LIV1A
Drug: Trastuzumab — Trastuzumab will be given by IV every 3 weeks at a dose of 6 mg/kg (the first dose will be 8 mg/kg)
  Other Names: Herceptin
  Arms: LV + Trastuzumab

SUMMARY:
This study will examine the safety and tolerability of ladiratuzumab vedotin (LV) in patients with metastatic breast cancer. LV will be given alone or in combination with trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of breast cancer with radiographic evidence of incurable, unresectable, locally advanced or metastatic disease (LA/MBC)
* One of the following:

  * Part A: Triple-negative disease (ER/PR/HER2-negative) and received at least 2 prior cytotoxic regimens in the incurable, unresectable, LA/MBC setting; or ER-positive and/or PR-positive/HER2-negative disease and received at least 2 prior cytotoxic regimens in the incurable, unresectable, LA/MBC setting and are no longer a candidate for hormonal therapy (not enrolling new patients);
  * Part B: Combination Arm: HER2-positive disease and received at least 2 prior cytotoxic regimens in the incurable, unresectable, LA/MBC setting (not enrolling new patients);
  * Part C: Triple-negative disease and received 2-4 prior non-hormonally-directed therapies in the MBC setting (not enrolling new patients);
  * Part D and Part E (dose-expansion cohort): Triple-negative disease and received 1 prior non-hormonally-directed or cytotoxic therapy in the MBC setting; or
  * Part E: HR+(ER-positive and/or PR-positive)/HER2-negative disease who are chemotherapy-eligible and not considered a candidate for further hormonal therapy. Must have received no more than 1 prior non-hormonally-directed or cytotoxic therapy in the LA/MBC setting.
* Part F: All of the following:

  * Triple negative breast cancer
  * No prior cytotoxic chemotherapy for unresectable locally advanced or metastatic stage disease
  * Tumor tissue PD-L1 expression CPS <10 expression
* Parts A, B, C, and D: Newly obtained or archived tumor tissue biopsy, must be collected for central pathology determination of LIV-1 expression
* Parts E and F: Archival or fresh baseline tumor sample is required.
* Measurable disease
* Eastern Cooperative Oncology Group performance status 0 or 1
* Combination Arm: adequate heart function

Exclusion Criteria:

* Pre-existing neuropathy Grade 2 or higher
* Parts A, B, C, and D: Cerebral/meningeal disease that is related to the underlying malignancy and has not been definitively treated. Parts E and F: Known or suspected cerebral/meningeal metastasis that has not been definitively treated.
* Prior treatment with LV or prior treatment with an MMAE-containing therapy
* Combination Arm: hypersensitivity to trastuzumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-02-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 1 month following last dose; up to approximately 2 years
  An AE is any untoward medical occurrence in a patient or clinical investigational subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Incidence of laboratory abnormalities | Through 1 month following last dose; up to approximately 2 years
  To be summarized using descriptive statistics.
Incidence of dose-limiting toxicity (DLT) | Through 3 weeks after first dose

SECONDARY OUTCOMES:
Blood concentrations of LV and metabolites | Through 3 weeks after dosing; up to approximately 2 years
Incidence of antitherapeutic antibodies | Through 1 month following last dose; up to approximately 2 years
Objective response rate (ORR) | Through 1 month following last dose; up to approximately 2 years
  ORR is defined as the proportion of patients with complete response (CR) or partial response (PR) per RECIST v1.1.
Duration of response (DOR) | Up to approximately 3 years
  DOR is defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression (clinical progression or progressive disease (PD) per RECIST v1.1).
Progression-free survival (PFS) | Up to approximately 8 years
  PFS is defined as the time from start of study treatment to first documentation of tumor progression (clinical progression or PD per RECIST v1.1).
Overall survival (OS) | Up to approximately 8 years
  OS is defined as the time from start of study treatment to date of death due to any cause.
PFS relative to prior therapy | Up to approximately 8 years
  The PFS ratio is defined for each subject as the ratio of the current PFS and the PFS achieved on their most recent therapy where they experienced progression.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Croft, PharmD, Study Director — Seagen Inc.; Zejing Wang, MD, PhD, Study Director — Seagen Inc.
Locations (38):
- United States (38):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - UC San Diego / Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center / Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - UCLA Medical Center / David Geffen School of Medicine, Santa Monica, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Poudre Valley Health System (PVHS), Fort Collins, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - The Whittingham Cancer Center / Norwalk Hospital, Norwalk, Connecticut
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University in St Louis, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Wake Forest Baptist Medical Center / Wake Forest University, Winston-Salem, North Carolina
  - Case Western Reserve University / University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Tennessee Oncology-Nashville/Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - Cancer Care Centers of South Texas - HOAST/Texas Oncology, New Braunfels, Texas
  - Northwest Medical Specialties, Puyallup, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia